CLINICAL TRIAL: NCT00131378
Title: Growth Hormone, Cardiovascular Risk, and Visceral Adiposity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Karen Klahr Miller, MD, Associate Professor of Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 525; MGH GCRC 678; 2004-P-000013; R01HL077674 (NIH)
Record Dates: First submitted 2005-08-16; First posted 2005-08-18 (Estimated); Results first posted 2014-03-06 (Estimated); Last update posted 2016-03-11 (Estimated); Status verified 2016-03

CONDITIONS: Obesity
Keywords: Visceral obesity; Growth hormone; Cardiovascular risk; Insulin resistance
MeSH Terms: conditions — Obesity; Obesity, Abdominal; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Male on GH (Experimental): Participants received growth hormone replacement therapy. The starting dose was 2 micrograms/kg per day and they were titrated within the normal range based on blood levels.
  Nutropin AQ growth hormone : Participants gave themselves injections of growth hormone every night for 6 months.
  Interventions: Drug: Nutropin AQ growth hormone
- Male on Placebo (Placebo Comparator): Participants received placebo.
  Placebo Growth Hormone : Participants gave themselves injections of placebo every night for 6 months.
  Interventions: Drug: Placebo Growth Hormone
- Female on GH (Experimental): Participants received growth hormone replacement therapy. The starting dose was 4 micrograms/kg per day and they were titrated within the normal range based on blood levels.
  Nutropin AQ growth hormone : Participants gave themselves injections of growth hormone every night for 6 months.
  Interventions: Drug: Nutropin AQ growth hormone
- Female on Placebo (Placebo Comparator): Participants received placebo.
  Placebo Growth Hormone : Participants gave themselves injections of placebo every night for 6 months.
  Interventions: Drug: Placebo Growth Hormone

INTERVENTIONS:
Drug: Nutropin AQ growth hormone — Participants will give themselves injections of growth hormone every night for 6 months.
  Arms: Female on GH; Male on GH
Drug: Placebo Growth Hormone — Participants will give themselves injections of placebo growth hormone every night for 6 months.
  Arms: Female on Placebo; Male on Placebo

SUMMARY:
This study will compare growth hormone levels and cardiovascular risk markers in normal weight and overweight women and men. In women and men with increased abdominal weight, growth hormone (GH) versus placebo will be administered and effects on cardiovascular risk, insulin resistance and body composition will be measured.

DETAILED DESCRIPTION:
The purpose of this study is to measure growth hormone levels in women and men who are normal weight, overweight, and obese. Growth hormone levels will be correlated with body weight, body composition, and markers of cardiovascular risk. In overweight or obese women and men with increased visceral adiposity and below average IGF-1 levels, growth hormone versus placebo will be given for 6 months. Effects of growth hormone treatment on weight, body composition, insulin resistance, lipids, and cardiovascular risk markers will then be assessed. Study subjects will be followed for an additional six months for these endpoints.

ELIGIBILITY:
Inclusion Criteria:

* For growth hormone measurement part (for men and women):

  1. For visceral adiposity arm: waist circumference greater than or equal to 88 cm for women or 102 cm for men, and BMI greater than or equal to 25 kg/m2
  2. For lean controls: BMI 18.5 to 24.9 kg/m2
* For growth hormone treatment part (for men and women):

  1. Visceral adiposity (waist circumference greater than or equal to 88 cm for women and 102 for men, BMI greater than or equal to 25 kg/m2)
  2. IGF-I within the lowest 2 quartiles for age and gender
  3. Willingness to maintain current activity level and diet

Exclusion Criteria:

* Diabetes mellitus (fasting plasma glucose greater than 126 mg/dL or 2-hour post-oral glucose tolerance test [OGTT] plasma glucose greater than 200)
* Taking the following medications in the last 3 months: weight loss or lipid-lowering agents, medications to treat diabetes mellitus or "pre-diabetes", oral contraceptives or estrogen-containing medications, other medications known to significantly affect weight
* Smoking
* Hematocrit below the lower limit of normal
* Amenorrhea for 3 months (in women)
* Pregnant or breastfeeding (in women)
* Polycystic ovary syndrome (in women)
* Weight that exceeds 280 pounds
* SGPT greater than 2 times the upper limit of normal
* History of malignancy, except for fully resolved basal cell carcinomas of the skin (Specific Aim 2 only)
* Radiation exposure greater than 1000 mrem over the last 12 months
* Previous diagnosis of cardiovascular disease
* History of pituitary or hypothalamic disease, brain radiation, or childhood growth hormone deficiency
* History of carpal tunnel syndrome that has not been surgically treated

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 142 (Actual)
Dates: Start 2004-11; Primary Completion 2012-11 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen K. Miller, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Dichtel LE, Bjerre M, Schorr M, Bredella MA, Gerweck AV, Russell BM, Frystyk J, Miller KK. The effect of growth hormone on bioactive IGF in overweight/obese women. Growth Horm IGF Res. 2018 Jun;40:20-27. doi: 10.1016/j.ghir.2018.03.003. Epub 2018 Mar 10. PMID 29679919
- [Derived] Bredella MA, Karastergiou K, Bos SA, Gerweck AV, Torriani M, Fried SK, Miller KK. GH administration decreases subcutaneous abdominal adipocyte size in men with abdominal obesity. Growth Horm IGF Res. 2017 Aug;35:17-20. doi: 10.1016/j.ghir.2017.06.001. Epub 2017 Jun 12. PMID 28628810
- [Derived] Bove RM, White CC, Gerweck AV, Mancuso SM, Bredella MA, Sherman JC, Miller KK. Effect of growth hormone on cognitive function in young women with abdominal obesity. Clin Endocrinol (Oxf). 2016 Apr;84(4):635-7. doi: 10.1111/cen.12996. Epub 2016 Feb 2. No abstract available. PMID 26663235
- [Derived] Dichtel LE, Yuen KC, Bredella MA, Gerweck AV, Russell BM, Riccio AD, Gurel MH, Sluss PM, Biller BM, Miller KK. Overweight/Obese adults with pituitary disorders require lower peak growth hormone cutoff values on glucagon stimulation testing to avoid overdiagnosis of growth hormone deficiency. J Clin Endocrinol Metab. 2014 Dec;99(12):4712-9. doi: 10.1210/jc.2014-2830. PMID 25210883
- [Derived] Bredella MA, Gerweck AV, Barber LA, Breggia A, Rosen CJ, Torriani M, Miller KK. Effects of growth hormone administration for 6 months on bone turnover and bone marrow fat in obese premenopausal women. Bone. 2014 May;62:29-35. doi: 10.1016/j.bone.2014.01.022. Epub 2014 Feb 5. PMID 24508386
- [Derived] Lin E, Bredella MA, Gerweck AV, Landa M, Schoenfeld D, Utz AL, Miller KK. Effects of growth hormone withdrawal in obese premenopausal women. Clin Endocrinol (Oxf). 2013 Jun;78(6):914-9. doi: 10.1111/cen.12102. PMID 23146135
- [Derived] Bredella MA, Lin E, Brick DJ, Gerweck AV, Harrington LM, Torriani M, Thomas BJ, Schoenfeld DA, Breggia A, Rosen CJ, Hemphill LC, Wu Z, Rifai N, Utz AL, Miller KK. Effects of GH in women with abdominal adiposity: a 6-month randomized, double-blind, placebo-controlled trial. Eur J Endocrinol. 2012 Apr;166(4):601-11. doi: 10.1530/EJE-11-1068. Epub 2012 Jan 24. PMID 22275471

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Female on GH | Female on Placebo | Male on GH | Male on Placebo
Started | 40 | 40 | 32 | 30
Completed | 29 | 22 | 22 | 21
Not Completed | 11 | 18 | 10 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Female on GH | Female on Placebo | Male on GH | Male on Placebo | Total
Number analyzed (Participants) | 40 | 40 | 32 | 30 | 142
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 40 | 40 | 32 | 30 | 142
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.7 (1.1) | 36.1 (1.1) | 32.4 (1.2) | 34.3 (1.1) | 34.6 (1.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 40 | 0 | 0 | 80
  Male | 0 | 0 | 32 | 30 | 62
Region of Enrollment [Number; unit: participants]
  United States | 40 | 40 | 32 | 30 | 142

OUTCOME MEASURES:

1. Primary Outcome: HsCRP
Description: 6 month change in HsCRP (primary cardiovascular risk endpoint)
Time Frame: Measured at baseline and month 6
Population: ITT
Measure: Mean (Standard Error); unit: mg/L
Arm/Group | Male on GH | Male on Placebo | Female on GH | Female on Placebo
Number analyzed (Participants) | 32 | 30 | 40 | 40
mg/L | -1.1 (0.5) | 0.5 (0.3) | -1.3 (0.2) | -0.3 (0.2)

2. Secondary Outcome: Measure of Insulin Resistance
Description: 6 month change in 2-hour glucose (primary insulin resistance endpoint)
Time Frame: Measured at baseline and month 6
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Male on GH | Male on Placebo | Female on GH | Female on Placebo
Number analyzed (Participants) | 32 | 30 | 40 | 40
mg/dL | 5.3 (5.6) | -12.5 (5.8) | 18.6 (6.3) | -0.9 (8.2)

3. Secondary Outcome: Insulin-like Growth Factor-1 (IGF-1) Levels
Description: 6-month change in IGF-1 levels
Time Frame: Measured at baseline and month 6
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Male on GH | Male on Placebo | Female on GH | Female on Placebo
Number analyzed (Participants) | 32 | 30 | 40 | 40
ng/mL | 179.0 (31.5) | 9.9 (7.8) | 106.5 (17.5) | -20.8 (7.6)

4. Primary Outcome: Total Abdominal Fat
Description: 6 month change in total abdominal fat (primary body composition endpoint)
Time Frame: Measured at baseline and month 6
Measure: Mean (Standard Error); unit: cm^2
Arm/Group | Female on GH | Female on Placebo
Number analyzed (Participants) | 40 | 40
cm^2 | -28.0 (9.7) | 1.5 (11)

5. Primary Outcome: Abdominal Fat
Description: 6 month change in visceral abdominal fat (primary body composition endpoint)
Time Frame: Measured at baseline and month 6
Measure: Mean (Standard Error); unit: cm^2
Arm/Group | Male on GH | Male on Placebo
Number analyzed (Participants) | 32 | 30
cm^2 | -15.9 (6.3) | -0.2 (7.2)

ADVERSE EVENTS:
Arm/Group | Female on GH | Female on Placebo | Male on GH | Male on Placebo
Serious Adverse Events (participants affected / at risk) | 0/40 | 1/40 | 0/32 | 1/30
Other Adverse Events (participants affected / at risk) | 4/40 | 3/40 | 7/32 | 3/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Female on GH (N=40) | Female on Placebo (N=40) | Male on GH (N=32) | Male on Placebo (N=30)
Breast Cancer (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Development of breast cancer in a subject on placebo.
MVA - motor vehicle accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Motor vehicle accident in a male subject on placebo.
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Female on GH (N=40) | Female on Placebo (N=40) | Male on GH (N=32) | Male on Placebo (N=30)
Abnormal Glucose Measurements (Endocrine disorders) | 2 (2) | 0 (0) | 4 (4) | 1 (1)
Carpel Tunnel Symptoms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Breast Calcification on Mammogram (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cervical HPV (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Goiter (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast Lump (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
New onset atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No